CLINICAL TRIAL: NCT00114829
Title: Preoperative Assessment of Colon Tumor: A Prospective, Blinded Study.
Brief Title: Preoperative Assessment of Colon Tumor
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Herlev Hospital (Other)
Collaborators: University Hospital, Gentofte, Copenhagen (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: Double | Purpose: Diagnostic
Other Study IDs: KA05028-MA; KA05028
Record Dates: First submitted 2005-06-17; First posted 2005-06-20 (Estimated); Last update posted 2006-03-09 (Estimated); Status verified 2005-05

CONDITIONS: Colorectal Cancer; Colorectal Tumor
Keywords: Colorectal cancer; Colorectal tumor; Dynamic contrast uptake; MR colonography
MeSH Terms: conditions — Colorectal Neoplasms

INTERVENTIONS:
Procedure: MR colonography with dynamic contrast uptake

SUMMARY:
The purpose of this study is to determine whether a colonic tumor can be classified as malignant or benign with magnetic resonance (MR) colonography. Patients with a verified colon carcinoma or benign tumor based on diverticulitis are offered a MR colonography with intravenous (I.V.) contrast. The tumor is classified as malignant or benign by assessing the dynamic contrast uptake and morphology. The Investigator is blinded from the verified diagnosis and the MR classification is compared to the histological diagnosis.

ELIGIBILITY:
Inclusion Criteria:

* Colorectal cancer
* Colorectal tumor

Exclusion Criteria:

* Active diverticulitis
* Pacemaker
* Metal in the body
* Claustrophobia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60
Dates: Start 2005-07

PRIMARY OUTCOMES:
Sensitivity in determining malignant or benign diagnose

SECONDARY OUTCOMES:
Sensitivity/specificity of MR colonography

CONTACTS AND LOCATIONS:
Overall Officials: Michael P Achiam, M.D., Principal Investigator — Department of Radiology Copenhagen University Hospital Herlev
Locations (1):
- Department of Radiology Copenhagen University Hospital Herlev, Herlev, Denmark

REFERENCES:
- [Derived] Achiam MP, Andersen LP, Klein M, Logager V, Chabanova E, Thomsen HS, Rosenberg J. Differentiation between benign and malignant colon tumors using fast dynamic gadolinium-enhanced MR colonography; a feasibility study. Eur J Radiol. 2010 Jun;74(3):e45-50. doi: 10.1016/j.ejrad.2009.03.033. Epub 2009 May 5. PMID 19419830